CLINICAL TRIAL: NCT01979120
Title: Validation of the "ApneaScan" Algorithm for the Detection of Sleep Disordered Breathing in Patients With Stable Symptomatic Chronic Heart Failure
Brief Title: Validation of the "ApneaScan" Algorithm for the Detection of Sleep Disordered Breathing in Chronic Heart Failure
Acronym: VASA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Christoph Schukro (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Dr. Christoph Schukro, Principle Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: ISROTH20033
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-08

CONDITIONS: Sleep-disordered Breathing; Chronic Heart Failure
Keywords: Sleep-disordered breathing; Chronic heart failure; Implantable cardioverter-defibrillator; Apnea-Hypopnea-Index; Portable Polygraphy Monitoring; Polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- only 1 cohort!: All patients already got an ICD implanted which includes an algorithm for screening of sleep-disordered breathing and will be examined by an portable polygraphy monitor in order to compare the Apnea-Hypopnea-Index.

SUMMARY:
A prospective observational multi-centre study for the validation of the ApneaScan algorithm (integrated in ICD devices (with or without cardiac resynchronization therapy function) of the "Incepta" series for the screening of sleep disordered breathing in patients with stable symptomatic chronic heart failure, using portable polygraphy monitoring device ("Embletta Gold") as reference for the Apnea-Hypopnea-Index (AHI).

Secondary objectives are the detection of severe sleep disordered breathing in patients with clinically indicated in-laboratory polysomnography, as well as correlations of the AHI detected by ApneaScan with other clinical endpoints like mortality, hospitalization, atrial fibrillation and ventricular arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patient´s written informed consent
* Patients with a cardiac rhythm management device (ICD with or without cardiac resynchronization therapy function) of the "Incepta" series (including the ApneaScan algorithm) already implanted for at least 8 weeks (corresponding to the duration of the leads´ healing process); in order to standardize the enrollment period, inclusion should be effected between the first (the earliest 8 weeks after implantation) and the second routine control of ICD-function (the latest 9 months after implantation)
* Stable symptomatic chronic heart failure for either ischemic or non-ischemic reason (moderately to severely impaired systolic left ventricular function with NYHA-class II to III) under optimal pharmacological treatment (according to guidelines 2012 of the European Society of Cardiology)

Exclusion Criteria:

* Unstable heart failure (NYHA-class IV) or asymptomatic chronic heart failure (including patients with very mild exercise induced dyspnea, i.e. NYHA-class I)
* Patients already treated for sleep apnea syndrome (i.e. continuous positive airway pressure mask) or chronic obstructive pulmonary disease with GOLD-class IV (i.e. long-term oxygen therapy)
* A limited AHI detection by the ApneaScan algorithm until the planned inclusion (randomly defined by <50% of countable AHI detection-points within the last 2 weeks).
* Patients with limited mobility due to orthopedic, neurologic or oncologic diseases (because of restricted assessment of exercise induced dyspnea)
* Patients on dialysis (either acute or chronic)
* Alcoholism or regular intake of hypnotics
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable symptomatic chronic heart failure and implanted ICD/CRT-D of the "INCEPTA" series
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea-Index | 1 night

SECONDARY OUTCOMES:
Apnea-Hypopnea-Index >/= 30 (in-laboratory polysomnography) | 1 night

OTHER OUTCOMES:
Mortality | 2 years
Hospitalization | 2 years
ICD therapies (i.e. shock or anti-tachycardia pacing) | 2 years
atrial fibrillation | 2 years
routine B-type natriuretic peptide | 1 night
  only if applicable!

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Schukro, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (14):
- Austria (5):
  - Hietzing Hospital, Vienna
  - Medical University of Vienna, Vienna
  - SMZO, Vienna
  - Wilhelminenspital, Vienna
  - Wiener Neustadt Hospital, Wiener Neustadt
- Germany (4):
  - Heart and Diabetes centre NRW, Bad Oeynhausen
  - Klinikum Coburg, Coburg
  - University of Leipzig, Leipzig
  - Reinbek Hospital, Reinbek
- Japan (4):
  - Kyushu University, Kyushu
  - Tokyo Medical University, Tokyo
  - Tottori University, Tottori
  - Juntendo University School of Medicine, Urayasu
- University of Geneva, Geneva, Switzerland